CLINICAL TRIAL: NCT03418376
Title: The Impact of Carnosine Loading and Rehabilitation Therapy on Exercise Capacity in Multiple Sclerosis.
Brief Title: Carnosine Loading and Periodized Training in MS and HC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Bert Op't Eijnde, Prof.Dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 17.09/REVA17.02
Record Dates: First submitted 2018-01-09; First posted 2018-02-01 (Actual); Results first posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Multiple Sclerosis; Exercise Therapy; Dietary Supplement
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Twenty multiple sclerosis (MS) patients and twenty healthy controls (HC), aged >18y will be included following written informed consent. Subjects will be excluded if they experience contraindications to participate in moderate to high intensity exercise or have an EDSS score >3. First, exercise capacity (maximal graded exercise test) will be evaluated. Heart function will be assessed by an experienced medical doctor, followed by measurement of body composition (DEXA). Maximal strength of the back- and abdominal muscles will be assessed to evaluate core stability. MS patients and HC will be randomly allocated to one of four intervention groups following 6 months of moderate-to-high-intensity cardiovascular exercise therapy with (MSβ, n=10; HCβ, n=10) or without (MSpla, n=10; HCplac, n=10) β-alanine supplementation. Groups not receiving β-alanine supplements, will receive placebo tablets. Following 6 months of exercise training (POST) measurements will be performed similar to baseline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All parties are blinded regarding the dietary supplement (beta-alanine) or placebo.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MS beta-alanine supplementation (Experimental): Subjects will perform a 6-month exercise intervention and receive beta-alanine supplements.
  Interventions: Dietary Supplement: Beta-alanine supplementation; Other: Exercise intervention
- MS placebo group (Placebo Comparator): Subjects will perform a 6-month exercise intervention and receive placebo tablets.
  Interventions: Other: Exercise intervention
- HC beta-alanine supplementation (Experimental): Subjects will perform a 6-month exercise intervention and receive beta-alanine supplements.
  Interventions: Dietary Supplement: Beta-alanine supplementation; Other: Exercise intervention
- HC placebo group (Placebo Comparator): Subjects will perform a 6-month exercise intervention and receive placebo tablets.
  Interventions: Other: Exercise intervention

INTERVENTIONS:
Dietary Supplement: Beta-alanine supplementation — The supplementation protocol of β-alanine (Etixx® Omega Pharma Belgium NV) involves oral intake of 4 x 800mg (3.2g/day29, 43) daily with at least 2h apart of slow-release β-alanine during the first 12 weeks. After this loading period, subjects will receive a maintenance dose of 2 x 800mg (1.6g/day) β-alanine for the remaining study duration.
  Arms: HC beta-alanine supplementation; MS beta-alanine supplementation
Other: Exercise intervention — The exercise training program (6 months) involves 3 week cycles (week I-III). During week I, subjects will perform high volume moderate intensity cardiovascular cycle training (3x/week). Twice a week, subjects perform 3h training sessions (70-80% HRmax*) and once a week a 1.5h session will be executed (80-90% HRmax). During week II, subjects will perform low volume maximum intensity interval cycle training (3/w). High intensity interval cycle training (HIIT) will consist of 3x maximal sprints (90-100% HRmax) of 1.5min, interspersed with 3min rest intervals. A 5min standardized warming up and 5min cooling down will be performed. Week III involves a recovery week where subjects will perform one training session of 1.5h at an exercise intensity of 70-80% HRmax and one session of HIIT.

SUMMARY:
Increasing evidence favours exercise therapy as an efficient tool to counteract inactivity related secondary symptoms in MS. Furthermore, exercise therapy may affect MS-associated muscle contractile and energy supply dysfunctions. So far, low to moderate intensity exercise rehabilitation has shown to induce small but consistent improvements in several functional parameters. High intensity exercise training in MS seems to further improve this. However, although results are promising, impairments in both muscle contraction and energy supply probably attenuate therapy outcome. In keeping with the above described physiological role of skeletal muscle carnosine and because muscle carnosine content may be lower in MS, the primary aim of the present project is to investigate whether carnosine loading improves exercise therapy outcome (exercise capacity, body composition) and performance in MS. If the latter hypothesis can be confirmed, muscle carnosine loading could be a novel intervention to improve exercise capacity and muscle function in this population.

DETAILED DESCRIPTION:
Pilot data from the (co-)applicants' laboratories suggest that EAE rats (animal MS model) and MS-patients suffer from significantly reduced muscle carnosine levels compared to healthy counterparts. The potential of β-alanine supplementation to elevate muscle carnosine content has been shown in healthy volunteers. Furthermore, the investigators have recently investigated β-alanine and carnosine supplementation in EAE animals. In MS, this has not been investigated yet. Therefore, the researchers' next step is to investigate the impact of β-alanine intake on exercise performance in MS patients. The investigators hypothesize that oral β-alanine supplementation improves exercise therapy outcomes in MS patients.

So far, it is clear that β-alanine intake enhances exercise capacity of untrained, trained and aged individuals by improving contractile properties, maintaining higher intracellular energy levels and optimizing training adaptations. Because early fatigue of contracting musculature during rehabilitation is the predominant cause of exercise cessation, postponing exercise-induced fatigue by β-alanine supplementation will be clinically very relevant (improving exercise therapy efficiency). Consequently, the investigators aim to research the ergogenic potential of β-alanine intake in MS rehabilitation and hypothesize that β-alanine supplementation optimizes exercise therapy outcome (exercise capacity, muscle contractile characteristics) in this population.

ELIGIBILITY:
Inclusion criteria:

Diagnosis Multiple Sclerosis. Healthy control. Aged >18y. Written informed consent.

Exclusion criteria:

Contraindications to perform moderate to high intensity exercise. Participation in another study. Experienced acute MS related exacerbation <6 months prior to start of the study EDSS score > 3.5

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bert O Eijnde, Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Diepenbeek, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MS Beta-alanine Supplementation; HC Beta-alanine Supplementation: Subjects will perform a 6-month intervention and receive beta-alanine supplements.
  Beta-alanine supplementation: The supplementation protocol of β-alanine (Etixx® Omega Pharma Belgium NV) involves oral intake of 4 x 800mg (3.2g/day29, 43) daily with at least 2h apart of slow-release β-alanine during the first 12 weeks. After this loading period, subjects will receive a maintenance dose of 2 x 800mg (1.6g/day) β-alanine for the remaining study duration.
  Exercise intervention: The exercise training program (6 months) involves 3 week cycles (week I-III). During week I, subjects will perform high volume moderate intensity cardiovascular cycle training (3x/week). Twice a week, subjects perform 3h training sessions (70-80% HRmax*) and once a week a 1.5h session will be executed (80-90% HRmax). During week II, subjects will perform low volume maximum intensity interval cycle training (3/w). High intensity interval cycle training (HIIT) will consist of 3x maximal sprints (90-100
Period: Overall Study
Arm/Group | MS Beta-alanine Supplementation | MS Placebo Group | HC Beta-alanine Supplementation | HC Placebo Group
Started | 12 | 11 | 11 | 11
Completed | 11 | 6 | 8 | 10
Not Completed | 1 | 5 | 3 | 1
Not completed — Musculoskeletal injury | 1 | 2 | 1 | 0
Not completed — Personal reasons | 0 | 2 | 2 | 1
Not completed — Exacerbation | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MS Beta-alanine Supplementation | MS Placebo Group | HC Beta-alanine Supplementation | HC Placebo Group | Total
Number analyzed (Participants) | 11 | 6 | 8 | 10 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (9.2) | 44 (5) | 43.3 (7.5) | 41.1 (11.7) | 42.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 1 | 5 | 12
  Male | 7 | 4 | 7 | 5 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 11 | 6 | 8 | 10 | 35
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 11 | 6 | 8 | 10 | 35

OUTCOME MEASURES:

1. Primary Outcome: VO2max
Description: Exercise capacity will be assessed using a maximal (12-lead ECG) graded cardiopulmonary exercise test (♂: 30W+15W/min, ♀: 20W+10W/min, GE eBike Basic®) with pulmonary gas exchange analysis (Jaeger Oxycon®). VO2max (maximal oxygen uptake) will be monitored. This test will be performed at least 48 hours separated from the muscle strength test, to prevent interference of muscle fatigue. Respiratory exchange ratio (RER) values will be evaluated to verify if the test was performed maximally (RER >1.1).
Time Frame: Before and after 6 months training (pre vs post)
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | MS Beta-alanine Supplementation | MS Placebo Group | HC Beta-alanine Supplementation | HC Placebo Group
Number analyzed (Participants) | 11 | 6 | 8 | 10
ml/kg/min | 40.4 (6.5) | 41.2 (7.9) | 44 (8.7) | 43.4 (8.6)

2. Primary Outcome: Serum Lactate
Description: During the exercise test, 2min capillary blood samples will be obtained to analyse blood lactate concentrations (Analox®) and determine the anaerobic threshold before, during and after exercise. Lactate max levels are the maximal concentrations measured during the test, whilst peak Lactate are the lactate concentrations following 2 minutes of rest after cessation of the maximal exercise test.
Time Frame: Before and after 6 months training (pre vs post)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MS Beta-alanine Supplementation | MS Placebo Group | HC Beta-alanine Supplementation | HC Placebo Group
Number analyzed (Participants) | 11 | 6 | 8 | 10
mmol/L
  Lactate max | 4.6 (2.0) | 4.4 (0.4) | 5.0 (1.2) | 5.1 (0.9)
  Lactate peak | 8.5 (2.6) | 9.2 (1.0) | 10.6 (2.6) | 8.9 (2.3)

3. Primary Outcome: Body Composition
Description: Whole body fat and lean tissue mass will be obtained using Dual Energy X-ray Absorptiometry scan (DEXA) (Hologic Series Delphi-A Fan Beam X-ray Bone Densitometer, Vilvoorde, Belgium). A calibrated analogue weight balance (Seca®) will be used to measure total body mass.
Time Frame: Before and after 6 months training (pre vs post)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | MS Beta-alanine Supplementation | MS Placebo Group | HC Beta-alanine Supplementation | HC Placebo Group
Number analyzed (Participants) | 11 | 6 | 8 | 10
kg
  Lean mss | 51.4 (7.0) | 49.2 (8.4) | 55.7 (7.7) | 50.3 (10.8)
  Fat mass | 16.8 (9.7) | 15.5 (6.6) | 14.6 (5.8) | 16.5 (5.2)

4. Primary Outcome: Strength Assessment Core Musculature
Description: Back- and abdominal muscle strength will be assessed using an isokinetic dynamometer (System 3, Biodex, ENRAF-NONIUS, New York, USA). After adequate warming-up and movement familiarization, subjects will perform 3 maximal isometric contractions of back- and abdominal muscles for 4-5sec. The peak value of the 3 maximal contractions will be reported (peak back, and peak abdominal muscles).
Time Frame: Before and after 6 months training (pre vs post)
Measure: Mean (Standard Deviation); unit: Nm
Arm/Group | MS Beta-alanine Supplementation | MS Placebo Group | HC Beta-alanine Supplementation | HC Placebo Group
Number analyzed (Participants) | 11 | 6 | 8 | 10
Nm
  Back | 257.4 (66.2) | 243.3 (80.3) | 243.5 (54.4) | 256 (87.7)
  Abdomen | 132.7 (28.9) | 145.3 (42.8) | 141 (35.9) | 149.5 (46.6)

5. Primary Outcome: Workload
Description: as for outcome 1
Time Frame: Before and after 6 months training (pre vs post)
Measure: Mean (Standard Deviation); unit: Wattage
Arm/Group | MS Beta-alanine Supplementation | MS Placebo Group | HC Beta-alanine Supplementation | HC Placebo Group
Number analyzed (Participants) | 11 | 6 | 8 | 10
Wattage | 209 (45) | 212 (41) | 248 (44) | 235 (59)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were not systematically assessed and reported. However, through personal communication with the participants, we have seen no adverse events. This was however not reported or assessed objectively.
  Adverse events were described as events that harmed the subjects as a consequence of the training/supplementation intervention.
Arm/Group | MS Beta-alanine Supplementation | MS Placebo Group | HC Beta-alanine Supplementation | HC Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT03418376/Prot_SAP_000.pdf
  • Informed Consent Form (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT03418376/ICF_001.pdf